CLINICAL TRIAL: NCT03496714
Title: Fading Safety Behaviors in an Internet-Based Secondary Prevention for Posttraumatic Stress Disorder
Brief Title: Online Psychoeducation for the Prevention of PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made to develop different intervention
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-11-0001
Record Dates: First submitted 2018-03-22; First posted 2018-04-12 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Psychoeducation on Trauma Reactions; Psychoeducation on Safety Behaviors and How to Fade Them; Monitoring-only Control
Keywords: Posttraumatic stress disorder; Safety behaviors; Threat appraisal; Secondary prevention; Internet-based; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Immediately after baseline assessment, each participant will be automatically randomized into one of three study conditions. Randomization will be stratified based on number and severity of safety behaviors used and level of Acute Stress Disorder symptoms reported at baseline. Once randomized, participants in the two psychoeducation conditions will immediately receive psychoeducation materials, and all participants will receive rationale for their study condition, as specified above. All three conditions will complete the same schedule of assessments.
Who Masked: Participant
Masking Description: Participants will be told of the specifications only of the condition to which they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PSYED-T (Active Comparator): In PSYED-T (psychoeducation on trauma symptoms), participants will receive a psychoeducation handout and watch a related video on common reactions to trauma. Participants in this condition will also receive a rationale stating that both learning about the nature of trauma reactions and monitoring symptoms are important for preventing development of PTSD.
  Interventions: Behavioral: Psychoeducation on trauma reactions
- PSYED-T+SB (Experimental): Participants in PSYED-T+SB (Combined psychoeducation on trauma reactions and safety behaviors) will receive psychoeducation handouts and videos on the nature of trauma symptoms and the nature of safety behaviors and how to fade them. Participants in this condition will also receive a rationale stating that learning about the nature of trauma reactions and safety behaviors, learning to fade safety behaviors, and monitoring symptoms are important in the prevention of PTSD.
  Interventions: Behavioral: Psychoeducation on trauma reactions; Behavioral: Psychoeducation on safety behaviors
- Monitoring-only control (No Intervention): The third condition will be a monitoring-only control and thus will receive no psychoeducation information. Participants in the control condition will receive a rationale that monitoring symptoms is important in the prevention of PTSD development.

INTERVENTIONS:
Behavioral: Psychoeducation on trauma reactions — The psychoeducation handout and video on trauma symptoms will discuss reactions that are common after experiencing a trauma.
  Other Names: PSYED-T
  Arms: PSYED-T; PSYED-T+SB
Behavioral: Psychoeducation on safety behaviors — The psychoeducation handout and video on safety behaviors will discuss safety behaviors that are common in PTSD and tips for how to eliminate them.
  Other Names: PSYED-SB
  Arms: PSYED-T+SB

SUMMARY:
Research on decreasing safety behaviors in therapy has been restricted to treatments for other anxiety disorders and has not included PTSD. In order to address this gap and to develop a widely accessible, cost-effective prevention, an internet-based, three-arm randomized secondary PTSD prevention trial is proposed. Self-help psychoeducation on common reactions to trauma and eliminating safety behaviors will be employed for participants who have recently experienced a traumatic event. Participants will be randomized to receive (a) psychoeducation on trauma symptoms only, (b) combined psychoeducation on trauma symptoms and eliminating safety behaviors, or (c) monitoring only control. All participants will monitor safety behaviors and trauma symptoms weekly for eight weeks. Psychoeducation materials will be handouts and videos administered online via REDCap.

It is hypothesized that participants in both psychoeducation conditions will have a lower incidence of PTSD, threat appraisal, and safety behaviors than participants in the monitoring-only control. It is also hypothesized that participants who receive combined psychoeducation on trauma symptoms and fading safety behaviors will have a lower incidence of PTSD, threat appraisal, and safety behaviors at Weeks 4 and 8 than will participants who receive psychoeducation on trauma symptoms only or participants in the monitoring-only control. It is further hypothesized that the effects of combined psychoeducation on preventing PTSD and threat appraisal will be mediated by decreased use of safety behaviors. Finally, it is hypothesized that combined psychoeducation on trauma symptoms and fading safety behaviors will be more effective in preventing PTSD for participants with higher levels of safety behaviors or threat appraisal at baseline. If effective, this secondary prevention program could be distributed widely to people who have recently experienced a trauma to prevent their development of PTSD.

DETAILED DESCRIPTION:
Baseline Assessment Participants will first access the study online through web links posted to widely accessible websites such as Facebook, Reddit, and Craigslist, and through The University of Texas at Austin PSY 301 SONA pool. Participants will also be recruited through Amazon Mechanical Turk. Participants will provide informed consent and will complete eligibility criteria, which will take approximately 5 minutes. Participants who meet eligibility criteria will immediately complete a baseline assessment, which will take approximately 25 minutes, including a basic demographics questionnaire and a thorough assessment of psychopathology symptoms and safety behaviors.

Randomization Immediately after baseline assessment, each participant will be automatically randomized into one of three study conditions. Randomization will be stratified based on number and severity of safety behaviors used and level of Acute Stress Disorder symptoms reported at baseline. Once randomized, participants in the two psychoeducation conditions will immediately receive psychoeducation materials, and all participants will receive rationale for their study condition, as specified below. All three conditions will complete the same schedule of assessments.

Conditions

Condition 1: Psychoeducation on trauma symptoms (PSYED-T) In Condition 1, participants will receive view a psychoeducation handout and video on trauma symptoms. Participants in this condition will also receive a rationale stating that learning about the nature of trauma reactions as well as monitoring trauma reactions and safety behaviors are important for preventing development of PTSD.

Condition 2: Combined psychoeducation on trauma symptoms and fading safety behaviors (PSYED-T+SB) Participants in Condition 2 will receive view a psychoeducation handout and video on trauma symptoms and on safety behaviors and how to fade them. Participants in this condition will also receive a rationale stating that learning about the nature of trauma reactions, learning to eliminate safety behaviors, and monitoring trauma reactions and safety behaviors are important in the prevention of PTSD.

Because it is expected that the psychoeducational information provided in PSYED-T+SB condition to be beneficial to participants, all participants will receive this information upon completion of the study.

Condition 3: Monitoring-only control Condition 3 will be a monitoring-only control and thus will receive no psychoeducation handouts or videos. Participants in this condition will receive a rationale that monitoring trauma reactions and safety behaviors is important in the prevention of PTSD development.

Psychoeducation At baseline, participants will receive a web link to the psychoeducation materials via email. Participants will then be instructed to carefully read the handout and watch the video and encouraged to revisit the materials throughout the course of the study. Immediately following baseline exposure to psychoeducation materials, all participants will complete a short quiz applicable to the psychoeducation and/or monitoring involved in their condition in order to ensure comprehension of the materials. Reading the psychoeducation materials, watching the video(s), and completing the quiz is expected to take participants approximately 30 minutes.

Participants will have unlimited access to the handouts and videos through a web link for the entire course of the study. Using REDCap, researchers will monitor the number of times each participant accesses psychoeducation materials during the study.

Weekly Assessments All participants will complete weekly assessments of trauma symptoms, threat appraisal, and safety behavior. Compliance with self-monitoring will be controlled for in all analyses.

Weeks 4 and 8 Assessments At Week 4 and Week 8, participants will complete a comprehensive assessment of all primary and secondary outcomes. Because the timing of onset of PTSD is variable among patients (Frueh, Grubaugh, Yeager, & Magruder, 2009), PTSD diagnosis will be assessed at Week 4 and Week 8. The psychoeducation quiz will also be administered at Weeks 4 and 8 to assess for comprehension and retention of the psychoeducational information.

Phone Interview The PSSI-5 interview will also be conducted over the phone for any participants who screen positive for PTSD at Week 4 or Week 8 based on the PSSI-5 self-report scale. The PSSI-5 phone interview will take approximately 20 minutes at each administration and will be audio recorded in order to assess inter-rater reliability of PTSD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Have regular access to the internet and email for eight weeks
* Have experienced a Criterion A trauma within the past 30 days, as assessed by the Life Events Checklist for DSM-5 (LEC-5; Weathers et al., 2013a)

Exclusion Criteria:

* Psychotic symptoms within the past six months, as measured by Psychiatric Diagnostic Screening Questionnaire (PDSQ) psychosis subscale
* Current suicidal intent, as measured by Beck Depression Inventory (BDI-II) suicidality item
* Immediate risk to others
* Have experienced a traumatic brain injury or other serious neurocognitive impairment in the past six months.
* Prior history of PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptom Scale Self-Report for DSM-5 (PSS-SR-5) | Week 4
  PTSD diagnosis at Week 4 will be measured by the PTSD Symptom Scale Self-Report for DSM-5 (PSS-SR-5).
PTSD Symptom Scale Self-Report for DSM-5 (PSS-SR-5) | Week 8
  PTSD diagnosis at Week 8 will be measured by the PTSD Symptom Scale Self-Report for DSM-5 (PSS-SR-5).
PTSD Symptom Scale Interview for DSM-5 (PSSI-5) | Week 4
  PTSD diagnosis at Week 4 will be measured by the PTSD Symptom Scale Interview for DSM-5 (PSSI-5). Only participants who meet criteria for PTSD based on the PSS-SR-5 will be assessed.
PTSD Symptom Scale Interview for DSM-5 (PSSI-5) | Week 8
  PTSD diagnosis at Week 8 will be measured by the PTSD Symptom Scale Interview for DSM-5 (PSSI-5). Only participants who meet criteria for PTSD based on the PSS-SR-5 will be assessed.
PTSD Checklist for DSM-5 (PCL-5) | Weekly change between baseline and Week 8
  Level of PTSD symptoms will be measured by the PTSD Checklist for DSM-5 (PCL-5).
PTSD Safety Behavior Inventory (PSBI) | Weekly change between baseline and Week 8
  The number of safety behaviors used will be measured by the PTSD Safety Behavior Inventory (PSBI).
Posttraumatic Cognitions Inventory (PTCI) | Weekly change between baseline and Week 8
  Level of threat appraisal will be measured by the Posttraumatic Cognitions Inventory (PTCI).

SECONDARY OUTCOMES:
Life Events Checklist for DSM-5 (LEC-5) | Week 0
  Type and experience of trauma occurring in the past 30 days will be measured by the Life Events Checklist for DSM-5 (LEC-5). Participants must select that one of the listed events has "Happened to me" in order to be eligible for this study.
National Stressful Events Survey Acute Stress Disorder Short Scale (NSESSS-ASD). | Week 0
  Symptoms of Acute Stress Disorder as defined by the DSM-5 will be measured using the National Stressful Events Survey Acute Stress Disorder Short Scale (NSESSS-ASD).
Acute Stress Disorder Scale (ASDS) | Week 0
  Acute Stress Disorder as defined by the DSM-IV will be measured by the Acute Stress Disorder Scale (ASDS).
Peritraumatic Dissociative Experiences Questionnaire (PDEQ) | Week 0
  Dissociation during the traumatic event will be measured by the Peritraumatic Dissociative Experiences Questionnaire (PDEQ).
Credibility and Expectancy Questionnaire (CEQ) | Week 0
  Credibility and expectancy of the intervention will be measured by selected items of the Credibility and Expectancy Questionnaire (CEQ).
Trauma Coping Self-Efficacy scale (CSE-T) | Weekly change between baseline and Week 8
  Perceived ability to cope with trauma-related situations will be measured by the Trauma Coping Self-Efficacy scale (CSE-T)
Anxiety Sensitivity Index (ASI-3) | Week 0, Week 4, Week 8
  Anxiety sensitivity will be measured by the Anxiety Sensitivity Index (ASI-3).
Beck Depression Inventory (BDI-II) | Week 0, Week 4, Week 8
  Depression will be measured by the Beck Depression Inventory (BDI-II).
Alcohol Use Disorders Identification Test - Short Version (AUDIT-C) | Weekly change between baseline and Week 8
  Drinking behaviors will be assessed with the AUDIT-C.
Patient Health Questionnaire-9 (PHQ-9) | Weekly change between baseline and Week 8
  Depressive symptoms will be assessed with the PHQ-9
Generalized Anxiety Disorder 7-item scale (GAD-7) | Weekly change between baseline and Week 8
  Symptoms of generalized anxiety disorder will be assessed with the GAD-7

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Telch, PhD, Principal Investigator — The University of Texas at Austin

IPD SHARING:
Plan to Share IPD: Undecided